CLINICAL TRIAL: NCT01121575
Title: A Phase 1, Open-label, Dose Escalation Study To Evaluate Safety, Pharmacokinetics And Pharmacodynamics Of Combined Oral C-met/Alk Inhibitor (Pf-02341066) And Pan-her Inhibitor (Pf-00299804) In Patients With Advanced Non-small Cell Lung Cancer
Brief Title: A Study Of Combined C- MET Inhibitor And PAN-HER Inhibitor (PF-02341066 And PF-00299804) In Patients With Non- Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8081006
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Phase 1 acquired resistance to erlotinib or gefitinib cMET inhibitor EGFR inhibitor panHER inhibitor combination trial Crizotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib; dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): PF-02341066 AND PF-00299804: Patients will be treated with combined cMET inhibitor (PF-02341066) and panHER inhibitor (PF-00299804).
  Interventions: Drug: PF-02341066; Drug: PF-00299804
- Arm 2 (Experimental): PF-00299804 FOLLOWED BY COMBINED PF-02341066 AND PF-00299804: Patients will be treated with single agent panHER inhibitor (PF-00299804) until disease progression and then with the maximum tolerated combined dose of cMET inhibitor (PF-02341066) and panHER inhibitor (PF-00299804).
  Interventions: Drug: PF-02341066; Drug: PF-00299804

INTERVENTIONS:
Drug: PF-02341066 — Arm 1: The starting dose will be 200 mg by mouth, twice a day of PF 02341066 in tablet form The dose of each drug in the combination [PF-02341066 and PF-00299804] will be escalated or de-escalated until the maximum tolerated combined dose is reached. Patients will then be treated with the maximum tolerated combined dose.
  Other Names: cMET inhibitor
  Arms: Arm 1
Drug: PF-00299804 — Arm 1: The starting dose will be 30 mg by mouth once a day of PF-0029804 in tablet form. The dose of each drug in the combination [PF-02341066 and PF-00299804] will be escalated or de-escalated until the maximum tolerated combined dose is reached. Patients will then be treated with the maximum tolerated combined dose.
  Other Names: panHER inhibitor
  Arms: Arm 1
Drug: PF-02341066 — Arm 2: With progressive disease the maximum tolerated combined dose of PF-02341066 (given by mouth twice a day in tablet form) and PF-00299804 (given by mouth once a day in tablet form).
  Other Names: cMET inhibitor
  Arms: Arm 2
Drug: PF-00299804 — Arm 2: The dose of 45 mg by mouth once a day of PF-00299804 in tablet form until progressive disease and then the maximum tolerated combined dose of PF-02341066 (given by mouth twice a day in tablet form) and PF-00299804 (given by mouth once a day in tablet form).
  Other Names: panHER inhibitor
  Arms: Arm 2

SUMMARY:
Lung cancer tumors become resistant to the first generation epidermal growth factor receptor (EGFR) inhibitors erlotinib or gefitinib by changing and increasing the activity of two cell signaling pathways: the cMET pathway and the EGFR pathway. Both resistance mechanisms can occur at the same time, in the same patient and even in the same tumor. This study combines a second generation EGFR inhibitor and a cMET inhibitor to block both these pathways in order to overcome resistance and treat this disease.

ELIGIBILITY:
Inclusion Criteria:

* advanced non small cell lung cancer (dose escalation phase)
* acquired resistance to erlotinib or gefitinib (expansion phase)
* mandatory entrance biopsy (expansion phase)

Exclusion Criteria:

* interstitial lung disease
* unstable brain metastases
* leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (8):
  - Clinical Trials Office University of Colorado Hospital (CTO), Aurora, Colorado
  - DRUG SHIPMENT: University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Lions Eye Institute, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - CCR, National Cancer Institute, Bethesda, Maryland
  - Drug Shipment Only, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
- Peter MacCallum Cancer Centre, Division of Haematology and Medical Oncology, East Melbourne, Victoria, Australia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081006&StudyName=A%20Study%20Of%20Combined%20C-%20MET%20Inhibitor%20And%20PAN-HER%20Inhibitor%20%28PF-02341066%20And%20PF-00299804%29%20In%20Patients%20With%20Non-%20Small%20Cell%20Lung%20Can

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 1, multicenter, open-label, non-randomized study of combined oral crizotinib and oral dacomitinib in participants with advanced non-small cell lung cancer (NSCLC). The study consisted of a dose Escalation Phase and an Expansion Phase. The Expansion Phase consisted of Expansion Cohort 1 and 2 which ran concurrently.
Pre-assignment Details: A total of 70 participants were enrolled and received study treatment in the United States (3 centers) and Australia (1 center). 33 participants in Escalation Phase and 37 participants in Expansion Phase (25 participants in Cohort 1 and 12 participants in Cohort 2) received treatment. The last participant completed the study on 11 Feb 2014.
Groups:
- Crizotinib 200 mg BID/ Dacomitinib 30 mg QD: Participants enrolled in dose escalation phase received combined oral crizotinib 200 mg twice a day (BID) and oral dacomitinib 30 mg once daily (QD). The first cycle was for 28 days thereafter, each cycle was 21 days.
- Crizotinib 200 mg BID/ Dacomitinib 45 mg QD: Participants received combined oral crizotinib 200 mg BID and oral dacomitinib 45 mg QD. The first cycle was for 28 days thereafter, each cycle was 21 days.
- Crizotinib 250 mg BID/ Dacomitinib 30 mg QD: Participants received combined oral crizotinib 250 mg BID and oral dacomitinib 30 mg QD. The first cycle was for 28 days thereafter, each cycle was 21 days.
- Crizotinib 250 mg QD/ Dacomitinib 45 mg QD: Participants received combined oral crizotinib 250 mg BID and oral dacomitinib 45 mg QD. The first cycle was for 28 days thereafter, each cycle was 21 days.
- Expansion Cohort 1: Participants enrolled in expansion cohort 1 received combined oral crizotinib and oral dacomitinib on a continuous daily schedule of crizotinib 200 mg BID + dacomitinib 30 mg QD. Each cycle was 21 days. If there was unacceptable toxicity or tolerability the dose could be adjusted to a lower combined dose. Expansion Cohort 1 was designed to examine the safety of crizotinib and dacomitinib administered concomitantly in NSCLC participants with acquired resistance to erlotinib or gefitinib.
- Expansion Cohort 2: Participants were treated first with single agent dacomitinib at a dose determined by agreement between the investigator and the sponsor, and then, at progression, with combined maximum tolerated dose of crizotinib and dacomitinib (given orally on a continuous schedule in 21-day cycles of crizotinib 200 mg BID + dacomitinib 30 mg QD) as soon as feasible, and no later than 28 days after documentation of progressive disease. Expansion Cohort 2 used the same participant population as Expansion Cohort 1 and was designed to assess the clinical value of adding crizotinib to dacomitinib treatment after disease progression on dacomitinib alone.
Period: Overall Study
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD | Expansion Cohort 1 | Expansion Cohort 2
Started | 14 | 6 | 7 | 6 | 25 | 12
Treated | 14 | 6 | 7 | 6 | 25 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 6 | 7 | 6 | 25 | 12
Not completed — Participant Refused Further Follow-Up | 0 | 0 | 0 | 0 | 5 | 1
Not completed — Unspecified Reasons | 8 | 6 | 7 | 5 | 13 | 10
Not completed — Death | 6 | 0 | 0 | 1 | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Crizotinib 200 mg BID/ Dacomitinib 30 mg QD: Participants enrolled in dose escalation phase received combined oral crizotinib 200 mg BID and oral dacomitinib 30 mg QD. The first cycle was for 28 days thereafter, each cycle was 21 days.
- Total: Total of all reporting groups
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD | Expansion Cohort 1 | Expansion Cohort 2 | Total
Number analyzed (Participants) | 14 | 6 | 7 | 6 | 25 | 12 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (9.87) | 61.7 (7.53) | 54.7 (11.34) | 62.2 (13.61) | 61.8 (10.83) | 59.6 (11.74) | 59.1 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 2 | 16 | 9 | 43
  Male | 9 | 1 | 1 | 4 | 9 | 3 | 27

OUTCOME MEASURES:

1. Primary Outcome: Overview of Treatment-emergent All Causalities Adverse Events (AEs) in Escalation Phase
Description: AE was any untoward medical occurrence with study drug/ device in a trial participant. Serious adverse event (SAE) was an AE resulting in death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity, congenital anomaly. Treatment-emergent AEs were those with initial onset or that worsen in severity after the first dose of study medication. AEs were reported from signing of informed consent until 28 days after the last dose of study medication. SAEs were reported after this time frame if considered to be treatment related. The severity of AEs were graded by the investigator using National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) v.4.02 and was assessed as Grade 0: no change from normal or reference range; Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening or disabling; Grade 5: death related to AE. However the below table included Grade 3, 4, and 5 AEs.
Time Frame: Up to Maximum of treatment duration + 28 days for each participant (could be 295 days)
Population: The safety analysis population included all enrolled participants who had received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 14 | 6 | 7 | 6
participants
  Participants with AEs | 14 | 6 | 7 | 6
  Participants with Grade 3 or 4 AEs | 9 | 4 | 5 | 5
  Participants with Grade 5 AEs | 3 | 0 | 0 | 1
  Participants with SAEs | 6 | 2 | 1 | 4

2. Primary Outcome: Overview of Treatment-emergent All Causalities AEs in Expansion Phase
Description: AE was any untoward medical occurrence with study drug/ device in a trial participant. SAE was an AE resulting in death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity, congenital anomaly. Treatment-emergent AEs were those with initial onset or that worsen in severity after the first dose of study medication. AEs were reported from signing of informed consent until 28 days after the last dose of study medication. SAEs were reported after this time frame if considered to be treatment related. The severity of AEs were graded by the investigator using NCI CTCAE v.4.02 and was assessed as Grade 0: no change from normal or reference range; Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening or disabling; Grade 5: death related to AE. However the below table included Grade 3, 4, and 5 AEs.
Time Frame: Up to Maximum of treatment duration + 28 days for each participant (could be 295 days)
Population: The safety analysis population included all enrolled participants who had received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 25 | 12
Participants
  Participants with AEs | 22 | 11
  Participants with Grade 3 or 4 AEs | 12 | 8
  Participants with Grade 5 AEs | 3 | 2
  Participants with SAEs | 8 | 8

3. Primary Outcome: Overview of Treatment-emergent, Treatment-related AEs in Escalation Phase
Description: An AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. SAE was an AE resulting in death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity, congenital anomaly. Treatment-emergent AEs were those with initial onset or that worsen in severity after the first dose of study medication. AEs were reported from signing of informed consent until 28 days after the last dose of study medication. SAEs were reported after this time frame if considered to be treatment related. The severity of AEs were graded by the investigator using NCI CTCAE v.4.02 and was assessed as Grade 0: no change from normal or reference range; Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening or disabling; Grade 5: death related to AE. However the below table included Grade 3, 4, and 5 AEs.
Time Frame: Up to Maximum of treatment duration + 28 days for each participant (could be 295 days)
Population: The safety analysis population included all enrolled participants who had received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 14 | 6 | 7 | 6
participants
  Participants with treatment-related AEs | 14 | 6 | 7 | 6
  Participants with treatment-related Grade 3/ 4 AEs | 8 | 3 | 3 | 3
  Participants with treatment-related Grade 5 AEs | 0 | 0 | 0 | 0
  Participants with treatment-related SAEs | 1 | 2 | 0 | 1

4. Primary Outcome: Overview of Treatment-emergent, Treatment-related AEs in Expansion Phase
Description: as for outcome 3
Time Frame: Up to Maximum of treatment duration + 28 days for each participant (could be 295 days)
Population: The safety analysis population included all enrolled participants who had received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 25 | 12
Participants
  Participants with treatment-related AEs | 22 | 11
  Participants with treatment-related Grade 3/ 4 AEs | 7 | 6
  Participants with treatment-related Grade 5 AEs | 0 | 0
  Participants with treatment-related SAEs | 3 | 3

5. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in Escalation Phase
Description: DLTs were those AEs which occurred in Cycle 1 of treatment in Dose Escalation Phase which may be attributed to study drug [combined Crizotinib (PF-02341066) plus Dacomitinib (PF-00299804)] without a clear alternative explanation and despite the use of adequate/maximal medical intervention as dictated by local institutional clinical practices or the judgment of the investigator. The following events were considered DLTs (using CTCAE version 4.02);1. Grade ≥4 hematologic events. 2. Grade ≥3 non-hematological events (except Grade 3/4 asymptomatic hypophosphatemia and Grade 3/4 hyperuricemia without signs and symptoms of gout). Nausea, vomiting or diarrhea had to have persisted at Grade 3 or 4 despite maximal medical therapy. Grade 3 hypertension will be considered a DLT only if the event is unmanageable by standard approved pharmacologic agents or if the symptomatic sequelae are identified despite appropriate medical intervention.
Time Frame: Cycle 1 (4 weeks)
Population: The DLT evaluable population was defined as safety analysis (SA) participants in the Dose Escalation phase who did not have a major treatment deviation during the first cycle.
Measure: Number; unit: Participants
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 14 | 6 | 7 | 6
Participants
  Grade 3 Alanine aminotransferase increased | 0 | 1 | 0 | 0
  Grade 3 Diarrhoea | 0 | 1 | 0 | 0
  Grade 3 Mucosal inflammation | 0 | 0 | 1 | 0

6. Secondary Outcome: Number of Participants With Stable Disease and Stable Disease Duration in Escalation Phase
Description: If a participant had not achieved an objective response with confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) - 1.1 as determined by the investigators, relative to the response evaluable population, but remained stable for at least 6 weeks after first dose, then the best overall response for such a participant was considered as stable disease.
Time Frame: From objective response to date of progression or death due to any cause, whichever occurs first (up to post treatment follow-up as 28-35 days after last dose of study treatment)
Population: The response evaluable population included participants in safety analysis population who had an adequate Baseline tumor assessment.
Measure: Number; unit: Participants
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 14 | 6 | 7 | 6
Participants
  Stable Disease | 10 | 3 | 2 | 5
  0- < 3 months | 3 | 2 | 1 | 0
  3- < 6 months | 6 | 1 | 1 | 3
  6- < 9 months | 1 | 0 | 0 | 2

7. Secondary Outcome: Number of Participants With Stable Disease and Stable Disease Duration in Expansion Phase
Description: If a participant had not achieved an objective response with confirmed complete response (CR) or partial response (PR) according to RECIST (1.1) as determined by the investigators, relative to the response evaluable population, but remained stable for at least 6 weeks after first dose, then the best overall response for such a participant was considered as stable disease.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 22 | 12
Participants
  Stable Disease | 6 | 5
  0- < 3 months | 1 | 0
  3- < 6 months | 4 | 4
  6- < 9 months | 1 | 1

8. Secondary Outcome: Number of Participants With Objective Response Rate (ORR) in Escalation Phase
Description: ORR was defined as the percent of participants with CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) determined by study physicians, relative to the response evaluable population. Participants were considered non-responders until proven otherwise. Thus, participants who: 1) Did not have CR or PR while on study, or 2) Did not have a post-baseline tumor evaluation, or 3) Received anti-tumor treatment other than the study medication prior to reaching a CR or PR, or 4) Died, in progress, or drop out for any reason prior to reaching a CR or PR, were counted as non-responders in the assessment of ORR. To be assigned a status of PR or CR, changes in tumor measurements in participants with responding tumors were confirmed by repeated tumor assessment that were performed 4 weeks after the criteria for response were first met.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 14 | 6 | 7 | 6
Participants | 0 [0.0 to 23.2] | 0 [0.0 to 45.9] | 0 [0.0 to 41.0] | 0 [0.0 to 45.9]

9. Secondary Outcome: Number of Participants With ORR in Expansion Phase
Description: as for outcome 8
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 22 | 12
Participants | 1 [0.1 to 22.8] | 0 [0.0 to 26.5]

10. Secondary Outcome: Duration of Response for the Only Participant Shown Partial Response in Expansion Phase
Description: This outcome measure presented the duration of response for one participant in expansion cohort 1 who showed partial response.
Time Frame: as for outcome 6
Population: This Outcome Measure was only assessed for participants with response.
Measure: Number; unit: Weeks
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 1 | 0
Weeks | 6.29 |

11. Secondary Outcome: Progression Free Survival (PFS) in Escalation Phase
Description: PFS was defined as the time from the date of the first dose to the date of the first documentation of objective tumor progression according to RECIST 1.1 or death on study due to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used.
Time Frame: From randomization to objective tumor progression or death (up to post treatment follow-up as 28-35 days after last dose of study treatment)
Population: The safety analysis population included all enrolled participants who had received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 14 | 6 | 7 | 6
Months | 3.1 [1.6 to 5.5] | 3.0 [1.5 to 4.4] | 1.7 [1.6 to 4.6] | 4.4 [1.6 to 7.2]

12. Secondary Outcome: Progression Free Survival (PFS) in Expansion Phase
Description: as for outcome 11
Time Frame: as for outcome 11
Population: The safety analysis population included all enrolled participants who had received at least 1 dose of study medication. In Expansion Cohort 1, two participants had censored reasons of "no adequate baseline", of which one participant had a censored reason "no tumor assessment data available.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 23 | 12
Months | 2.1 [1.4 to 4.4] | 2.1 [1.4 to 5.3]

13. Secondary Outcome: Expression Analysis of Tumor Biomarkers (HGF, EGFR, and c-Met ) at Baseline Using Immunohistochemistry (IHC) Method
Description: Tumor biomarkers such as HGF, EGFR, and c-Met were analyzed in tumor cells (neoplastic compartment) of tumor specimens from both expansion cohorts 1 and 2 by IHC. The H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+, where 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum calculated score of 0 to maximum calculated score of 300, where 0 correspond to no expression and maximum score of 300 indicates the strongest expression. However, the biomarker expression level (higher or lower) was not a predictor of outcome.
Time Frame: Baseline
Population: The tumor analysis population included participants in safety analysis population who had a screening and on-treatment tumor biopsy for assessment of tumor biomarkers.
Measure: Median (Full Range); unit: H-Score
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 23 | 12
H-Score
  HGF (N= 19, 11) | 40.0 [0 to 280] | 67.0 [0 to 104]
  EGFR (N= 14, 8) | 193.2 [2 to 300] | 170.0 [7 to 300]
  cMet (N= 19, 11) | 125.0 [0 to 300] | 165.0 [20 to 299]

14. Secondary Outcome: Expression Analysis of Tumor Biomarkers (EGFR, and c-Met) at Baseline Using Fluorescent in Situ Hybridization (FISH) Method
Description: Expression of tumor biomarkers EGFR and cMet at Baseline (using FISH method) are presented in this outcome measure.
Time Frame: Baseline
Population: as for outcome 13
Measure: Median (Full Range); unit: Ratio
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 23 | 12
Ratio
  Ratio of Red to Green of EGFR (N= 11, 11) | 1.580 [0.98 to 3.59] | 1.180 [0.94 to 4.63]
  Ratio of Green to Orange for cMET (N = 19, 11) | 1.040 [0.43 to 2.12] | 1.000 [0.88 to 1.10]

15. Secondary Outcome: Number of Participants With c-Met, HER2, EGFR Amplification and ALK Rearrangement at Baseline Using FISH Method
Description: Participants showed amplification of c-Met, HER2, and EGFR in the tumor cells and gene rearrangement of ALK are presented in this outcome measure.
Time Frame: Baseline
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 23 | 12
Participants
  c-Met amplification (N= 19, 11) | 1 [0.98 to 3.59] | 0 [0.94 to 4.63]
  HER2 amplification (N= 19, 7) | 0 | 0
  EGFR amplification (N= 11,11) | 2 | 3
  ALK rearrangement (N= 19, 11) | 0 | 0

16. Secondary Outcome: Plasma Concentration of sMet by Study Visits
Description: This outcome measure presented the plasma concentration of sMet at different study visits. s-Met was analyzed using an enzyme-linked immunosorbent assay (ELISA).
Time Frame: At screening and Cycle 1 Day 1 (C1D1) (6 hours post dose), and C1D15, C2D1, C2D15 (all predose).
Population: The soluble protein analysis population included participants in safety analysis who had a screening or C1D1 soluble protein assessment, and at least one on-treatment soluble protein assessment (C1D14 C2D1 or C2D14).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 21 | 7
pg/mL
  Baseline at Screening | 1353411.8 (349746.88) [2.67 to 10.40] | 1557000.0 (514352.02) [2.05 to 25.20]
  C1D1 | 1519047.6 (230995.77) | 1450500.0 (553557.13)
  C1D15 | 1483157.9 (243904.64) | 1676666.7 (540246.86)
  C2D1 | 1525666.7 (394836.61) | 1540000.0 (315515.45)
  C2D15 | 1564666.7 (224367.90) | 1602500.0 (126589.89)

17. Secondary Outcome: Number of Participants With EGFR Mutation at Baseline
Description: Sample analyses were performed in accordance to Good Laboratory Practice (GLP) guidance and included mutation detection for EGFR gene.
Time Frame: Baseline
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 23 | 12
Participants
  Exon 18 (G719X) | 1 | 1
  Exon 19 (Deletion) | 6 | 3
  Exon 20 (T790M) | 6 | 3
  Exon 20 (T790M/S768I) | 1 | 0
  Exon 20 (S768I) | 0 | 1
  Exon 21 (L858R) | 6 | 1

18. Secondary Outcome: Number of Participants With KRAS Mutation (GLY12CYS) at Baseline
Description: Sample analyses were performed in accordance to GLP guidance and included mutation detection for KRAS gene.
Time Frame: Baseline
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 23 | 12
Participants | 1 | 0

19. Secondary Outcome: Number of Participants With PIK3CA Mutation at Baseline
Description: Sample analyses were performed in accordance to GLP guidance and included mutation detection for PIK3CA gene.
Time Frame: Baseline
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 23 | 12
Participants
  Exon 20 (M1004I) (N= 14, 6) | 1 | 0
  Exon 20 (Q1061K) (N= 14, 6) | 1 | 0
  Exon 20 (H1047R) (N= 14, 6) | 2 | 0
  Exon 9 (E545K) (N= 14, 6) | 1 | 0

20. Secondary Outcome: Number of Participants With ROS1 Gene Translocation at Baseline
Description: Sample analyses were performed in accordance to GLP guidance and included translocation detection (RNA based) for ROS1 gene.
Time Frame: Baseline
Population: The tumor analysis population included participants in safety analysis population who had a screening and on-treatment tumor biopsy for assessment of tumor biomarkers. However, number of participants analyzed in the below table included the participants evaluated for ROS1 gene translocation.
Measure: Number; unit: Participants
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

21. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Escalation Phase - Area Under the Plasma Concentration-time Profile From Time Zero to the Last Quantifiable Concentration (AUClast)
Description: At each designated time point, blood samples (3 mL) for pharmacokinetic (PK) analysis of crizotinib and its metabolite, PF 06260182 were collected in appropriately labeled collection tubes containing dipotassium ethylenediamine tetra-acetic acid (K2EDTA). The below analysis table included AUClast for crizotinib and PF-06260182. AUClast was calculated using Linear/Log trapezoidal method.
Time Frame: Cycle 1 (C1)/Day 1 (D1), C1D15
Population: The PK parameter analysis population was defined as all participants in the safety analysis population who had at least 1 of the PK parameters of interest. N= Number of participants in the treatment group in the indicated population. n= Number of participants contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 11 | 6 | 7 | 6
ng•hr/mL
  Crizotinib C1D1 - single dose (n= 11, 6, 7, 6) | 509.7 (62) | 420.8 (53) | 506.6 (29) | 656.6 (65)
  Crizotinib C1D15 multiple dose (n=8, 3, 6, 5) | 1759 (39) | 2464 (14) | 1732 (35) | 1672 (44)
  PF-06260182 C1D1 - single dose (n= 11, 6, 7, 6) | 121.3 (76) | 103.2 (74) | 121.6 (29) | 220.7 (55)
  PF-06260182 C1D15 - multiple dose (n=8, 3, 6, 5) | 382.3 (52) | 593.5 (53) | 440.5 (37) | 532.0 (68)

22. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Escalation Phase - Area Under the Plasma Concentration-time Curve 10 (AUC10)
Description: At each designated time point, blood samples (3 mL) for pharmacokinetic (PK) analysis of crizotinib and its metabolite, PF 06260182 were collected in appropriately labeled collection tubes containing dipotassium ethylenediamine tetra-acetic acid (K2EDTA). AUC10 was calculated using Linear/Log trapezoidal method. The below analysis table included geometric Mean and Geometric Coefficient of Variation of AUC10 for crizotinib and PF-06260182. Arithmetic mean was presented if the n=2.
Time Frame: C1D1, C1D15
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 11 | 6 | 7 | 6
ng•hr/mL
  Crizotinib C1D1 - single dose (n= 8, 3, 4, 6) | 624.9 (57) | 500.8 (9) | 559.6 (26) | 655.8 (65)
  Crizotinib C1D15 multiple dose (n= 5, 2, 6, 5) | 2000 (43) | 2620 (NA) — Not applicable as arithmetic mean is presented for n = 2. | 1732 (35) | 1644 (44)
  PF-06260182 C1D1 - single dose (n= 8, 3, 4, 6) | 162.1 (57) | 127.6 (32) | 141.5 (25) | 228.0 (57)
  PF-06260182 C1D15 - multiple dose (n= 5, 2, 6, 5) | 452.5 (48) | 798.0 (NA) — Not applicable as arithmetic mean is presented for n = 2. | 473.3 (39) | 525.5 (68)

23. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Escalation Phase - Maximum Plasma Concentration (Cmax)
Description: At each designated time point, blood samples (3 mL) for pharmacokinetic (PK) analysis of crizotinib and its metabolite, PF 06260182 were collected in appropriately labeled collection tubes containing dipotassium ethylenediamine tetra-acetic acid (K2EDTA). The below analysis table included Cmax for crizotinib and PF-06260182. Cmax was observed directly from data.
Time Frame: C1D1, C1D15
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 11 | 6 | 7 | 6
ng/mL
  Crizotinib C1D1 - single dose (n= 11, 6, 7, 6) | 84.24 (58) | 94.13 (22) | 90.86 (29) | 114.0 (61)
  Crizotinib C1D15 multiple dose (n=8, 3, 6, 5) | 231.5 (41) | 329.7 (12) | 218.1 (33) | 268.9 (77)
  PF-06260182 C1D1 - single dose (n= 11, 6, 7, 6) | 18.50 (72) | 22.37 (26) | 20.97 (29) | 34.33 (61)
  PF-06260182 C1D15 - multiple dose (n=8, 3, 6, 5) | 49.73 (50) | 78.45 (44) | 57.56 (34) | 83.23 (91)

24. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Escalation Phase - Time of Last Quantifiable Concentration (Tlast)
Description: At each designated time point, blood samples (3 mL) for pharmacokinetic (PK) analysis of crizotinib and its metabolite, PF 06260182 were collected in appropriately labeled collection tubes containing dipotassium ethylenediamine tetra-acetic acid (K2EDTA). The below analysis table included Tlast for crizotinib and PF-06260182. Tlast was observed directly from data.
Time Frame: C1D1, C1D15
Population: as for outcome 21
Measure: Median (Full Range); unit: Hour
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 11 | 6 | 7 | 6
Hour
  Crizotinib C1D1 - single dose (n= 11, 6, 7, 6) | 9.92 (58) [7.83 to 10.1] | 9.33 (22) [4.08 to 10.0] | 9.05 (29) [7.55 to 9.95] | 9.75 (61) [9.00 to 10.2]
  Crizotinib C1D15 multiple dose (n=8, 3, 6, 5) | 9.29 (41) [7.62 to 9.98] | 9.42 (25) [8.00 to 9.92] | 9.05 (47) [9.00 to 9.57] | 10.2 (35) [10.0 to 10.5]
  PF-06260182 C1D1 - single dose (n= 11, 6, 7, 6) | 9.92 (72) [7.83 to 10.1] | 9.33 (26) [4.08 to 10.0] | 9.05 (29) [7.55 to 9.95] | 9.75 (61) [9.00 to 10.2]
  PF-06260182 C1D15 - multiple dose (n=8, 3, 6, 5) | 9.29 (50) [7.62 to 9.98] | 9.42 (44) [8.00 to 9.92] | 9.05 (34) [9.00 to 9.57] | 10.2 (91) [10.0 to 10.5]

25. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Escalation Phase -Time to Maximum Plasma Concentration (Tmax)
Description: At each designated time point, blood samples (3 mL) for pharmacokinetic (PK) analysis of crizotinib and its metabolite, PF 06260182 were collected in appropriately labeled collection tubes containing dipotassium ethylenediamine tetra-acetic acid (K2EDTA). The below analysis table included Tmax for crizotinib and PF-06260182. Tmax was observed directly from data as time of first occurrence.
Time Frame: C1D1, C1D15
Population: as for outcome 21
Measure: Median (Full Range); unit: Hour
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 11 | 6 | 7 | 6
Hour
  Crizotinib C1D1 - single dose (n= 11, 6, 7, 6) | 3.00 (58) [1.00 to 6.00] | 3.53 (22) [2.00 to 4.00] | 3.92 (29) [2.00 to 6.07] | 3.06 (61) [3.00 to 4.00]
  Crizotinib C1D15 multiple dose (n=8, 3, 6, 5) | 1.68 (41) [0.0 to 7.97] | 6.17 (25) [3.97 to 8.00] | 2.00 (47) [0.0 to 6.00] | 6.00 (35) [1.98 to 8.00]
  PF-06260182 C1D1 - single dose (n= 11, 6, 7, 6) | 4.07 (72) [3.00 to 8.00] | 4.00 (26) [3.02 to 6.05] | 3.98 (29) [3.00 to 6.07] | 4.99 (61) [3.03 to 6.10]
  PF-06260182 C1D15 - multiple dose (n=8, 3, 6, 5) | 4.03 (50) [0.0 to 7.97] | 6.17 (44) [3.97 to 8.00] | 4.09 (34) [3.00 to 6.02] | 6.00 (91) [4.02 to 6.05]

26. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Escalation Phase - AUClast
Description: At each designated time point, blood samples (3 mL) for PK analysis of dacomitinib and its metabolite, PF 05199265 were collected in appropriately labeled collection tubes containing dipotassium ethylenediamine tetra-acetic acid (K2EDTA). The below analysis table included AUClast for dacomitinib and PF-05199265. AUClast was calculated using Linear/Log trapezoidal method.
Time Frame: C1D1, C1D15
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 11 | 6 | 7 | 6
ng•hr/mL
  Dacomitinib C1D1 - single dose (n= 10, 6, 7, 5) | 208.3 (72) [1.00 to 6.00] | 132.3 (153) [2.00 to 4.00] | 146.3 (86) [2.00 to 6.07] | 307.7 (56) [3.00 to 4.00]
  Dacomitinib C1D15 multiple dose (n= 8, 4, 6, 4) | 1339 (47) [0.0 to 7.97] | 2343 (70) [3.97 to 8.00] | 1212 (15) [0.0 to 6.00] | 1775 (31) [1.98 to 8.00]
  PF-5199265 C1D1 - single dose (n= 8, 6, 6, 6) | 27.68 (80) [3.00 to 8.00] | 7.438 (115) [3.02 to 6.05] | 10.19 (190) [3.00 to 6.07] | 55.00 (75) [3.03 to 6.10]
  PF-06260182 C1D15 - multiple dose (n= 8, 4, 6, 4) | 51.48 (108) [0.0 to 7.97] | 52.24 (78) [3.97 to 8.00] | 44.97 (90) [3.00 to 6.02] | 161.0 (33) [4.02 to 6.05]

27. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Escalation Phase - AUC24
Description: At each designated time point, blood samples (3 mL) for PK analysis of dacomitinib and its metabolite, PF 05199265 were collected in appropriately labeled collection tubes containing dipotassium ethylenediamine tetra-acetic acid (K2EDTA). The below analysis table included AUC24 for dacomitinib and PF-05199265. AUC24 was calculated using Linear/Log trapezoidal method.
Time Frame: C1D1, C1D15
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 11 | 6 | 7 | 6
ng•hr/mL
  Dacomitinib C1D1 - single dose (n= 8, 3, 5, 5) | 252.7 (61) [1.00 to 6.00] | 347.9 (26) [2.00 to 4.00] | 223.4 (23) [2.00 to 6.07] | 306.6 (57) [3.00 to 4.00]
  Dacomitinib C1D15 multiple dose (n= 8, 4, 6, 4) | 1336 (48) [0.0 to 7.97] | 2334 (69) [3.97 to 8.00] | 1203 (15) [0.0 to 6.00] | 1745 (30) [1.98 to 8.00]
  PF-5199265 C1D1 - single dose (n= 9, 3, 5, 6) | 28.57 (87) [3.00 to 8.00] | 14.80 (51) [3.02 to 6.05] | 16.08 (169) [3.00 to 6.07] | 54.72 (76) [3.03 to 6.10]
  PF-06260182 C1D15 - multiple dose (n= 8, 4, 6, 4) | 51.37 (108) [0.0 to 7.97] | 51.97 (78) [3.97 to 8.00] | 44.72 (90) [3.00 to 6.02] | 158.1 (31) [4.02 to 6.05]

28. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Escalation Phase - Cmax
Description: At each designated time point, blood samples (3 mL) for PK analysis of dacomitinib and its metabolite, PF 05199265 were collected in appropriately labeled collection tubes containing dipotassium ethylenediamine tetra-acetic acid (K2EDTA). The below analysis table included Cmax for dacomitinib and PF-05199265. Cmax was observed directly from data.
Time Frame: C1D1, C1D15
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 11 | 6 | 7 | 6
ng/mL
  Dacomitinib C1D1 - single dose (n= 10, 6, 7, 5) | 15.56 (58) [1.00 to 6.00] | 17.49 (23) [2.00 to 4.00] | 12.40 (21) [2.00 to 6.07] | 18.22 (64) [3.00 to 4.00]
  Dacomitinib C1D15 multiple dose (n= 8, 4, 6, 4) | 65.00 (52) [0.0 to 7.97] | 122.4 (75) [3.97 to 8.00] | 57.04 (13) [0.0 to 6.00] | 86.81 (38) [1.98 to 8.00]
  PF-5199265 C1D1 - single dose (n= 10, 6, 6, 7) | 1.894 (89) [3.00 to 8.00] | 0.9888 (79) [3.02 to 6.05] | 0.8833 (130) [3.00 to 6.07] | 3.193 (74) [3.03 to 6.10]
  PF-06260182 C1D15 - multiple dose (n= 8, 4, 6, 4) | 2.367 (115) [0.0 to 7.97] | 2.649 (75) [3.97 to 8.00] | 2.073 (95) [3.00 to 6.02] | 7.560 (34) [4.02 to 6.05]

29. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Escalation Phase - Tlast
Description: At each designated time point, blood samples (3 mL) for PK analysis of dacomitinib and its metabolite, PF 05199265 were collected in appropriately labeled collection tubes containing dipotassium ethylenediamine tetra-acetic acid (K2EDTA). The below analysis table included Tlast for dacomitinib and PF-05199265. Tlast was observed directly from data.
Time Frame: C1D1, C1D15
Population: as for outcome 21
Measure: Median (Full Range); unit: Hour
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 11 | 6 | 7 | 6
Hour
  Dacomitinib C1D1 - single dose (n= 11, 6, 7, 5) | 24.0 (8.00) [8.00 to 24.6] | 15.9 (15.9) [4.08 to 24.0] | 23.6 (24.0) [7.55 to 24.1] | 24.0 [23.0 to 24.3]
  Dacomitinib C1D15 multiple dose (n= 8, 4, 6, 4) | 24.00 [23.0 to 24.3] | 23.9 [23.5 to 24.5] | 23.9 [22.9 to 24.8] | 24.4 [24.0 to 25.6]
  PF-5199265 C1D1 - single dose (n= 8, 6, 6, 6) | 24.0 [8.00 to 24.6] | 15.9 [4.08 to 24.0] | 23.5 [7.55 to 24.1] | 24.1 [23.0 to 24.5]
  PF-06260182 C1D15 - multiple dose (n= 8, 4, 6, 4) | 24.0 [23.0 to 24.3] | 23.9 [23.5 to 24.5] | 23.9 [22.9 to 24.8] | 24.4 [24.0 to 25.6]

30. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Escalation Phase - Tmax
Description: At each designated time point, blood samples (3 mL) for PK analysis of dacomitinib and its metabolite, PF 05199265 were collected in appropriately labeled collection tubes containing dipotassium ethylenediamine tetra-acetic acid (K2EDTA). The below analysis table included Tmax for dacomitinib and PF-05199265. Tmax was observed directly from data as time of first occurrence.
Time Frame: C1D1, C1D15
Population: as for outcome 21
Measure: Median (Full Range); unit: Hour
Arm/Group | Crizotinib 200 mg BID/ Dacomitinib 30 mg QD | Crizotinib 200 mg BID/ Dacomitinib 45 mg QD | Crizotinib 250 mg BID/ Dacomitinib 30 mg QD | Crizotinib 250 mg QD/ Dacomitinib 45 mg QD
Number analyzed (Participants) | 11 | 6 | 7 | 6
Hour
  Dacomitinib C1D1 - single dose (n= 11, 6, 7, 5) | 5.99 (8.00) [3.93 to 24.1] | 8.03 (15.9) [4.08 to 24.0] | 6.00 (24.0) [5.92 to 8.05] | 6.17 [5.92 to 8.00]
  Dacomitinib C1D15 multiple dose (n= 8, 4, 6, 4) | 6.00 [0.0 to 23.1] | 5.09 [3.97 to 23.5] | 6.09 [4.15 to 8.13] | 5.00 [4.00 to 6.00]
  PF-5199265 C1D1 - single dose (n= 8, 6, 6, 6) | 6.95 [3.93 to 24.1] | 4.04 [3.97 to 8.00] | 6.78 [3.98 to 8.05] | 6.08 [3.98 to 24.3]
  PF-06260182 C1D15 - multiple dose (n= 8, 4, 6, 4) | 6.98 [0.0 to 23.1] | 3.95 [2.00 to 6.17] | 5.92 [0.0 to 23.9] | 2.00 [0.0 to 5.98]

31. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Expansion Cohort 1 With or Without Co-administration of Dacomitinib - AUClast
Description: Participants were evaluated for the effect of dacomitinib on steady-state PK of crizotinib. PK of crizotinib alone was evaluated on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) after a lead in period of continuous BID dosing of crizotinib for approximately 12 days (±2 days). PK of crizotinib and dacomitinib in combination treatment was evaluated on Day 1 of Cycle 2. Blood samples for crizotinib full PK were to be collected on Day -1 and Day 1 of Cycle 2. The below table included PK data for AUClast. AUClast was calculated using Linear/Log trapezoidal method.
Time Frame: Day -1 (crizotinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Groups:
- Crizotinib Alone (Expansion Cohort 1): Participants received crizotinib alone continuous 200 mg BID dosing for approximately 12 days (±2 days).
- Crizotinib + Dacomitinib (Expansion Cohort 1): Participants received combined oral crizotinib (200 mg BID) and oral dacomitinib (30 mg QD) on a continuous daily schedule.
Arm/Group | Crizotinib Alone (Expansion Cohort 1) | Crizotinib + Dacomitinib (Expansion Cohort 1)
Number analyzed (Participants) | 19 | 19
ng•hr/mL
  Crizotinib (n = 16, 13) | 2223 (53) [3.93 to 24.6] | 1365 (47) [4.08 to 24.0]
  PF-06260182 (n = 16, 13) | 616.3 (77) | 356.6 (61)
Statistical Analysis 1: Comparison: Crizotinib Alone (Expansion Cohort 1) vs Crizotinib + Dacomitinib (Expansion Cohort 1); Statistical analysis was performed for crizotinib AUClast for participants who had both Day -1 and C2D1 data. Result for the analysis of AUClast was based on data from 11 participants. No statistical analysis was performed for PF-06260182; Test type: Superiority or Other; Ratio of adjust geometric mean = 69.25, 90% CI 2-sided [54.22 to 88.44] — Ratio of crizotinib + dacomitinib / crizotinib alone adjust geometric mean was analyzed using the mixed effect model and displayed as percentage

32. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Expansion Cohort 1 With or Without Co-administration of Dacomitinib - AUC10
Description: Participants were evaluated for the effect of dacomitinib on steady-state PK of crizotinib. PK of crizotinib alone was evaluated on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) after a lead in period of continuous BID dosing of crizotinib for approximately 12 days (±2 days). PK of crizotinib and dacomitinib in combination treatment was evaluated on Day 1 of Cycle 2. Blood samples for crizotinib full PK were to be collected on Day -1 and Day 1 of Cycle 2. The below table included PK data for AUC10. AUC10 was calculated using Linear/Log trapezoidal method.
Time Frame: Day -1 (crizotinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Groups:
- Crizotinib + Dacomitinib (Expansion Cohort 1): Participants received combined oral crizotinib (200 mg BID) and oral dacomitinib (30 mg QD) on a continuous daily schedule. Each cycle was 21 days.
Arm/Group | Crizotinib Alone (Expansion Cohort 1) | Crizotinib + Dacomitinib (Expansion Cohort 1)
Number analyzed (Participants) | 19 | 19
ng•hr/mL
  Crizotinib (n = 11, 9) | 2167 (56) [3.93 to 24.6] | 1489 (44) [4.08 to 24.0]
  PF-06260182 (n = 11, 9) | 634.3 (82) | 422.3 (55)
Statistical Analysis 1: Comparison: Crizotinib Alone (Expansion Cohort 1) vs Crizotinib + Dacomitinib (Expansion Cohort 1); Statistical analysis was performed for crizotinib AUC10 for participants who had both Day -1 and C2D1 data. Result for the analysis of AUC10 was based on data from 6 participants. No statistical analysis was performed for PF-06260182; Test type: Superiority or Other; Ratio of adjust geometric mean = 78.84, 90% CI 2-sided [58.90 to 105.54] — [estimate comment as in outcome 31, analysis 1]

33. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Expansion Cohort 1 With or Without Co-administration of Dacomitinib - Cmin
Description: Participants were evaluated for the effect of dacomitinib on steady-state PK of crizotinib. PK of crizotinib alone was evaluated on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) after a lead in period of continuous BID dosing of crizotinib for approximately 12 days (±2 days). PK of crizotinib and dacomitinib in combination treatment was evaluated on Day 1 of Cycle 2. Blood samples for crizotinib full PK were to be collected on Day -1 and Day 1 of Cycle 2. The below table included PK data for Cmin. Cmin was observed directly from data.
Time Frame: Day -1 (crizotinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Crizotinib Alone (Expansion Cohort 1) | Crizotinib + Dacomitinib (Expansion Cohort 1)
Number analyzed (Participants) | 19 | 19
ng/mL
  Crizotinib (n = 16, 13) | 181.8 (64) [3.93 to 24.6] | 102.8 (51) [4.08 to 24.0]
  PF-06260182 (n = 16, 13) | 47.22 (99) | 25.53 (60)

34. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Expansion Cohort 1 With or Without Co-administration of Dacomitinib - Cmax
Description: Participants were evaluated for the effect of dacomitinib on steady-state PK of crizotinib. PK of crizotinib alone was evaluated on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) after a lead in period of continuous BID dosing of crizotinib for approximately 12 days (±2 days). PK of crizotinib and dacomitinib in combination treatment was evaluated on Day 1 of Cycle 2. Blood samples for crizotinib full PK were to be collected on Day -1 and Day 1 of Cycle 2. The below table included PK data for Cmax. Cmax was observed directly from data.
Time Frame: Day -1 (crizotinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Crizotinib Alone (Expansion Cohort 1) | Crizotinib + Dacomitinib (Expansion Cohort 1)
Number analyzed (Participants) | 19 | 19
ng/mL
  Crizotinib (n = 16, 13) | 306.0 (57) [3.93 to 24.6] | 191.5 (43) [4.08 to 24.0]
  PF-06260182 (n = 16, 13) | 82.92 (79) | 51.15 (56)
Statistical Analysis 1: Comparison: Crizotinib Alone (Expansion Cohort 1) vs Crizotinib + Dacomitinib (Expansion Cohort 1); Statistical analysis was performed for crizotinib Cmax for participants who had both Day -1 and C2D1 data. Result for the analysis of Cmax was based on data from 11 participants. No statistical analysis was performed for PF-06260182; Test type: Superiority or Other; Ration of adjust geometric mean = 70.60, 90% CI 2-sided [54.71 to 91.12] — [estimate comment as in outcome 31, analysis 1]

35. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Expansion Cohort 1 With or Without Co-administration of Dacomitinib - Tlast
Description: Participants were evaluated for the effect of dacomitinib on steady-state PK of crizotinib. PK of crizotinib alone was evaluated on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) after a lead in period of continuous BID dosing of crizotinib for approximately 12 days (±2 days). PK of crizotinib and dacomitinib in combination treatment was evaluated on Day 1 of Cycle 2. Blood samples for crizotinib full PK were to be collected on Day -1 and Day 1 of Cycle 2. The below table included PK data for Tlast. Tlast was observed directly from data.
Time Frame: Day -1 (crizotinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Median (Full Range); unit: Hour
Arm/Group | Crizotinib Alone (Expansion Cohort 1) | Crizotinib + Dacomitinib (Expansion Cohort 1)
Number analyzed (Participants) | 19 | 19
Hour
  Crizotinib (n = 16, 13) | 9.650 (57) [7.63 to 10.1] | 9.000 (43) [7.67 to 10.0]
  PF-06260182 (n = 16, 13) | 9.650 (79) [7.63 to 10.1] | 9.000 (56) [7.67 to 10.0]

36. Secondary Outcome: Plasma Crizotinib and PF-06260182 Pharmacokinetic Parameter in Expansion Cohort 1 With or Without Co-administration of Dacomitinib - Tmax
Description: Participants were evaluated for the effect of dacomitinib on steady-state PK of crizotinib. PK of crizotinib alone was evaluated on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) after a lead in period of continuous BID dosing of crizotinib for approximately 12 days (±2 days). PK of crizotinib and dacomitinib in combination treatment was evaluated on Day 1 of Cycle 2. Blood samples for crizotinib full PK were to be collected on Day -1 and Day 1 of Cycle 2. The below table included PK data for Tmax. Tmax was observed directly from data as time of first occurrence.
Time Frame: Day -1 (crizotinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Median (Full Range); unit: Hour
Arm/Group | Crizotinib Alone (Expansion Cohort 1) | Crizotinib + Dacomitinib (Expansion Cohort 1)
Number analyzed (Participants) | 19 | 19
Hour
  Crizotinib (n = 16, 13) | 2.04 (57) [0.0 to 4.00] | 3.20 (43) [2.02 to 9.00]
  PF-06260182 (n = 16, 13) | 3.96 (79) [1.97 to 10.1] | 3.95 (56) [2.02 to 7.67]

37. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Expansion Cohort 2 With or Without Co-administration of Dacomitinib - AUClast
Description: PK samples for full PK evaluation of dacomitinib were drawn on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) and on C2D1. Dacomitinib and PF-05199265 PK parameter (AUClast) following dacomitinib alone and in combination with crizotinib are summarized in the below table. AUClast was calculated using Linear/Log trapezoidal method.
Time Frame: Day -1 (dacomitinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Groups:
- Dacomitinib Alone (Expansion Cohort 2): Participants received dacomitinib (30 mg, QD) alone in 21-day cycles until disease progression.
- Crizotinib + Dacomitinib (Expansion Cohort 2): Participants who progressed on dacomitinib were changed from single agent dacomitinib at the prevailing dose to combined maximum tolerated dose of crizotinib and dacomitinib (given orally on a continuous schedule in 21-day cycles) as soon as feasible, and no later than 28 days after documentation of disease progression. The participants in this group received 30 mg QD doses of dacomitinib in combination with 200 mg BID doses of crizotinib.
Arm/Group | Dacomitinib Alone (Expansion Cohort 2) | Crizotinib + Dacomitinib (Expansion Cohort 2)
Number analyzed (Participants) | 10 | 10
ng•hr/mL
  Dacomitinib (n = 6, 5) | 1016 (45) [0.0 to 4.00] | 1148 (44) [2.02 to 9.00]
  PF-05199265 (n = 7, 6) | 80.94 (598) [1.97 to 10.1] | 78.22 (42) [2.02 to 7.67]
Statistical Analysis 1: Comparison: Dacomitinib Alone (Expansion Cohort 2) vs Crizotinib + Dacomitinib (Expansion Cohort 2); Statistical analysis was performed for dacomitinib AUClast for participants who had both Day -1 and C2D1 data. Result for the analysis of AUClast was based on data from 3 participants. No statistical analysis was performed for PF-05199265; Test type: Superiority or Other; Ratio of adjust geometric mean = 117.81, 90% CI 2-sided [64.97 to 213.61] — Ratio of crizotinib + dacomitinib / dacomitinib alone adjust geometric mean was analyzed using the mixed effect model and displayed as percentage

38. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Expansion Cohort 2 With or Without Co-administration of Dacomitinib - AUC24
Description: PK samples for full PK evaluation of dacomitinib were drawn on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) and on C2D1. Dacomitinib and PF-05199265 PK parameter (AUC24) following dacomitinib alone and in combination with crizotinib are summarized in the below table. AUC24 was calculated using Linear/Log trapezoidal method.
Time Frame: Day -1 (dacomitinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Dacomitinib Alone (Expansion Cohort 2) | Crizotinib + Dacomitinib (Expansion Cohort 2)
Number analyzed (Participants) | 10 | 10
ng•hr/mL
  Dacomitinib (n = 6, 5) | 995.7 (45) [0.0 to 4.00] | 1148 (44) [2.02 to 9.00]
  PF-05199265 (n = 7, 6) | 78.57 (587) [1.97 to 10.1] | 78.36 (42) [2.02 to 7.67]
Statistical Analysis 1: Comparison: Dacomitinib Alone (Expansion Cohort 2) vs Crizotinib + Dacomitinib (Expansion Cohort 2); Statistical analysis was performed for dacomitinib AUC24 for participants who had both Day -1 and C2D1 data. Result for the analysis of AUC24 was based on data from 3 participants. No statistical analysis was performed for PF-05199265; Test type: Superiority or Other; Ratio of adjust geometric mean = 121.90, 90% CI 2-sided [70.20 to 211.66] — [estimate comment as in outcome 37, analysis 1]

39. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Expansion Cohort 2 With or Without Co-administration of Dacomitinib - Cmin
Description: PK samples for full PK evaluation of dacomitinib were drawn on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) and on C2D1. Dacomitinib and PF-05199265 PK parameter (Cmin) following dacomitinib alone and in combination with crizotinib are summarized in the below table. Cmin was observed directly from data.
Time Frame: Day -1 (dacomitinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dacomitinib Alone (Expansion Cohort 2) | Crizotinib + Dacomitinib (Expansion Cohort 2)
Number analyzed (Participants) | 10 | 10
ng/mL
  Dacomitinib (n = 6, 5) | 33.11 (58) [0.0 to 4.00] | 39.92 (47) [2.02 to 9.00]
  PF-05199265 (n = 7, 6) | 5.440 (83) [1.97 to 10.1] | 2.901 (47) [2.02 to 7.67]

40. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Expansion Cohort 2 With or Without Co-administration of Dacomitinib - Cmax
Description: PK samples for full PK evaluation of dacomitinib were drawn on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) and on C2D1. Dacomitinib and PF-05199265 PK parameter (Cmax) following dacomitinib alone and in combination with crizotinib are summarized in the below table. Cmax was observed directly from data.
Time Frame: Day -1 (dacomitinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dacomitinib Alone (Expansion Cohort 2) | Crizotinib + Dacomitinib (Expansion Cohort 2)
Number analyzed (Participants) | 10 | 10
ng/mL
  Dacomitinib (n = 6, 5) | 47.15 (44) [0.0 to 4.00] | 59.58 (49) [2.02 to 9.00]
  PF-05199265 (n = 7, 6) | 4.222 (375) [1.97 to 10.1] | 4.070 (37) [2.02 to 7.67]
Statistical Analysis 1: Comparison: Dacomitinib Alone (Expansion Cohort 2) vs Crizotinib + Dacomitinib (Expansion Cohort 2); Statistical analysis was performed for dacomitinib Cmax for participants who had both Day -1 and C2D1 data. Result for the analysis of Cmax was based on data from 3 participants. No statistical analysis was performed for PF-05199265; Test type: Superiority or Other; Ratio of adjust geometric mean = 130.57, 90% CI 2-sided [82.46 to 206.73] — [estimate comment as in outcome 37, analysis 1]

41. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Expansion Cohort 2 With or Without Co-administration of Dacomitinib - Tlast
Description: PK samples for full PK evaluation of dacomitinib were drawn on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) and on C2D1. Dacomitinib and PF-05199265 PK parameter (Tlast) following dacomitinib alone and in combination with crizotinib are summarized in the below table. Tlast was observed directly from data.
Time Frame: Day -1 (dacomitinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Median (Full Range); unit: Hour
Arm/Group | Dacomitinib Alone (Expansion Cohort 2) | Crizotinib + Dacomitinib (Expansion Cohort 2)
Number analyzed (Participants) | 10 | 10
Hour
  Dacomitinib (n = 6, 5) | 24.40 (44) [24.0 to 26.2] | 23.80 (49) [22.6 to 24.0]
  PF-05199265 (n = 7, 6) | 24.50 (375) [24.0 to 26.2] | 23.80 (37) [22.6 to 24.0]

42. Secondary Outcome: Plasma Dacomitinib and PF-05199265 Pharmacokinetic Parameter in Expansion Cohort 2 With or Without Co-administration of Dacomitinib - Tmax
Description: PK samples for full PK evaluation of dacomitinib were drawn on Day -1 (one day before C1D1 on which the combination treatment of crizotinib and dacomitinib started) and on C2D1. Dacomitinib and PF-05199265 PK parameter (Tmax) following dacomitinib alone and in combination with crizotinib are summarized in the below table. Tmax was observed directly from data as time of first occurrence.
Time Frame: Day -1 (dacomitinib alone), C2D1 (crizotinib + dacomitinib)
Population: as for outcome 21
Measure: Median (Full Range); unit: Hour
Arm/Group | Dacomitinib Alone (Expansion Cohort 2) | Crizotinib + Dacomitinib (Expansion Cohort 2)
Number analyzed (Participants) | 10 | 10
Hour
  Dacomitinib (n = 6, 5) | 16.0 (44) [5.90 to 24.6] | 5.92 (49) [3.83 to 9.80]
  PF-05199265 (n = 7, 6) | 5.90 (375) [0.0 to 25.5] | 4.35 (37) [0.0 to 23.8]

ADVERSE EVENTS:
Time Frame: Up to Maximum of treatment duration + 28 days for each participant (could be 295 days)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. The below tables included all causality SAEs (frequency threshold 0%) and AEs ( frequency threshold 5%).
Groups:
- PF-02341066, 200 mg BID/ PF-00299804, 30 mg QD: Participants enrolled in dose escalation phase received combined oral crizotinib 200 mg BID and oral dacomitinib 30 mg. The first cycle was for 28 days thereafter, each cycle was 21 days.
- PF-02341066, 200 mg BID/ PF-00299804, 45 mg QD: Participants enrolled in dose escalation received combined oral crizotinib 200 mg BID and oral dacomitinib 45 mg. The first cycle was for 28 days thereafter, each cycle was 21 days.
- PF-02341066, 250 mg BID/ PF-00299804, 30 mg QD: Participants enrolled in dose escalation received combined oral crizotinib 250 mg BID and oral dacomitinib 30 mg. The first cycle was for 28 days thereafter, each cycle was 21 days.
- PF-02341066, 250 mg QD/ PF-00299804, 45 mg QD: Participants enrolled in dose escalation received combined oral crizotinib 250 mg BID and oral dacomitinib 45 mg. The first cycle was for 28 days thereafter, each cycle was 21 days.
Arm/Group | PF-02341066, 200 mg BID/ PF-00299804, 30 mg QD | PF-02341066, 200 mg BID/ PF-00299804, 45 mg QD | PF-02341066, 250 mg BID/ PF-00299804, 30 mg QD | PF-02341066, 250 mg QD/ PF-00299804, 45 mg QD | Expansion Cohort 1 | Expansion Cohort 2
Serious Adverse Events (participants affected / at risk) | 6/14 | 2/6 | 1/7 | 4/6 | 9/25 | 9/12
Other Adverse Events (participants affected / at risk) | 14/14 | 6/6 | 7/7 | 6/6 | 25/25 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02341066, 200 mg BID/ PF-00299804, 30 mg QD (N=14) | PF-02341066, 200 mg BID/ PF-00299804, 45 mg QD (N=6) | PF-02341066, 250 mg BID/ PF-00299804, 30 mg QD (N=7) | PF-02341066, 250 mg QD/ PF-00299804, 45 mg QD (N=6) | Expansion Cohort 1 (N=25) | Expansion Cohort 2 (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 2 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02341066, 200 mg BID/ PF-00299804, 30 mg QD (N=14) | PF-02341066, 200 mg BID/ PF-00299804, 45 mg QD (N=6) | PF-02341066, 250 mg BID/ PF-00299804, 30 mg QD (N=7) | PF-02341066, 250 mg QD/ PF-00299804, 45 mg QD (N=6) | Expansion Cohort 1 (N=25) | Expansion Cohort 2 (N=12)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 1 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 3 | 0
Hypogonadism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 0 | 2 | 2
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eye inflammation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 1 | 0 | 0 | 4 | 0
Punctate keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pupils unequal (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Trichiasis (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 4 | 2 | 3 | 0 | 5 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Chapped lips (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 12 | 6 | 6 | 6 | 19 | 10
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 9 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 10 | 4 | 5 | 6 | 19 | 10
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rectal lesion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 4 | 2
Vomiting (Gastrointestinal disorders) | 9 | 2 | 1 | 5 | 11 | 6
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 1 | 0
Axillary pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 2 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 7 | 3 | 3 | 3 | 13 | 7
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 2 | 0
Local swelling (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 3 | 2 | 6 | 2
Oedema (General disorders) | 1 | 0 | 0 | 1 | 3 | 0
Oedema peripheral (General disorders) | 7 | 2 | 3 | 1 | 7 | 4
Pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Intertrigo candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Omphalitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 6 | 2 | 1 | 3 | 8 | 7
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 2 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Chemical eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0 | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 1 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1 | 1 | 2 | 2
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 3 | 0 | 0 | 0 | 2 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 4 | 3 | 3 | 10 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 4 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1 | 0 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 3 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 2 | 0 | 2 | 3 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 0 | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 1 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 3 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 0 | 2 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 3 | 10 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 2 | 1 | 3 | 6 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Facial wasting (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 3 | 3 | 3 | 5 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 3 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 2 | 0 | 1 | 1 | 2 | 0
Intra-abdominal haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Poor venous access (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites.

Investigator may not disclose previously undisclosed confidential information other than study results.